CLINICAL TRIAL: NCT00540189
Title: Initial Versus Delayed Operation for Treatment of Complicated Appendicitis In Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to adequatly recruit
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Steven W. Bruch, Clinical Assoicate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00007791
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Perforated Appendicitis
Keywords: appendicitis, perforated, children
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial appendectomy (Other): children with complicated appendicitis will undergo initial appendectomy
  Interventions: Procedure: Initial appendectomy
- Interval appendectomy (Other): children with complicated appendicitis will undergo initial antibiotic treatment followed by an interval appendectomy
  Interventions: Procedure: Interval appendectomy

INTERVENTIONS:
Procedure: Initial appendectomy
  Arms: Initial appendectomy
Procedure: Interval appendectomy
  Arms: Interval appendectomy

SUMMARY:
To determine the most cost effective way to treat children with perforated appendicitis we will randomize all children presenting with perforated appendicitis to initial operation, with in 24 hours of admission, or to initial antibiotics, with or without percutaneous drainage, and subsequent interval appendectomy after 8 weeks. Our outcomes will include cost, complications, length of stay, and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:children

* Age 2-17 with a diagnosis of perforated appendicitis

Exclusion Criteria:

* Age <2 and >18
* Pregnancy
* Immunocompromise

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
cost effectiveness | 3 months post entry into the study

CONTACTS AND LOCATIONS:
Overall Officials: Steven W Bruch, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- Mott Childrens Hospital, Ann Arbor, Michigan, United States